CLINICAL TRIAL: NCT07283029
Title: Evaluating Changes in Functional Fitness Following a 10-Week Home-Based Comprehensive Exercise Program in Endometrial Cancer Patients Who Have Completed Treatment
Brief Title: Activity and Cancer Survivorship Exercise Pilot
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Jess S. Gorzelitz, Assistant Professor, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 202212082
Record Dates: First submitted 2025-11-20; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Intervention (Experimental)
  Interventions: Other: Functional fitness following home-based comprehensive exercise program

INTERVENTIONS:
Other: Functional fitness following home-based comprehensive exercise program — Patients complete a home-based exercise program, receive remote health coaching sessions, and complete functional fitness tests on study. Patients also wear a Fitbit and receive health education on study.

SUMMARY:
This early phase I clinical trial measures the changes in functional fitness following home-based comprehensive exercise program in patients who have endometrial cancer who have completed treatment. Endometrial cancer is an increasingly common diagnosis, with health and quality of life concerns persisting after the active cancer treatment period. Exercise in cancer survivors has the potential to reduce the risk of death by improving cardiovascular fitness, quality of life, strength, longevity, and independence. A home-based exercise programs may be a feasible approach for exercise programming in patients who have endometrial cancer who have completed treatment.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide written informed consent
* Willing to comply with all study procedures and be available for the duration of the study
* Fluent in spoken and written English
* Women 18-74 years of age
* Documented diagnosis of type I, stage I-IIIc endometrial cancer within the past 5 years
* Completion of current treatment for endometrial cancer
* Technology access (cellphone with data, broadband internet, WiFi) for tele coaching
* Pass the Physical Activity Readiness Questionnaire (PAR-Q)

Exclusion Criteria:

* Absolute contraindications to exercise (i.e., acute myocardial infarction, severe orthopedic or musculoskeletal limitations
* Have evidence of recurrent or metastatic disease
* Are currently performing resistance training >= 2 days per week
* Are currently exceeding 150 minutes of at least moderate intensity activity per week
* Report of chest pain, shortness of breath, fainting, or angina pectoris
* Have physical disability that would limit range of motion through exercises such as sitting, standing and inability to walk one block
* Plans to move from the area
* Enrolled in another clinical trial or has used of any investigational drugs, biologics, or devices within 30 days prior to randomization
* Women who are pregnant or breast-feeding
* Not suitable for study participation due to other reasons at the discretion of the investigator
* Failing the Physical Activity Readiness Questionnaire

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Chair sit to stand test | baseline, pre-intervention and immediately after the intervention
  Will be assessed using the Functional Fitness Test, which is a battery of six tests including the 30 second chair stand, the 30 second arm curl, the 6-minute walk, the chair sit and reach, the 8-foot up and go, and the back scratch tests. Mixed effects regression models will be used to estimate changes in each of the 6 tests included in the Functional Fitness Test from pre- to post-intervention. Random effects will be included to account for the longitudinally correlated nature of repeat measurements within a patient. Estimated mean changes and associated 90% confidence intervals will be reported. Primary outcome is number of repetitions in the chair sit to stand test

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 10 weeks
  Will be summarized by system organ class and/or preferred term, type of adverse event, severity (based on National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, [NCI CTCAE v 5.0] grades), and relation to study treatment. The most severe grade per patient will be reported.
Muscle strengthening exercise session adherence | Up to 10 weeks
  Exercise session adherence will be defined as the proportion of planned exercise sessions in which a participant completes at least 50% of the prescribed exercises. The mean and associated 90% confidence interval will be reported
Aerobic physical activity adherence | Up to 10 weeks
  Aerobic physical activity adherence will be defined as the proportion of planned weeks a participant accumulates 150 minutes of moderate intensity activity. The mean and associated 90% confidence interval will be reported.
Tele coaching adherence | Up to 10 weeks
  Tele coaching adherence will be defined as the proportion of planned exercise sessions in which a participant completes. The mean and associated 90% confidence interval will be reported.
Exercise program acceptability | Up to 10 weeks
  Acceptability will be assessed using Likert scale ratings of quality of exercise equipment, educational materials, health coaching, study feedback and distance-delivery format. Means and associated 90% confidence intervals will be reported for each item.
Body weight | baseline, pre-intervention and immediately after the intervention
  Will be assessed by the within patient change of weight, waist and hip circumferences will be assessed from pre- to post-intervention. Mixed effects regression models will be used to estimate changes in anthropometrics. Random effects will be included to account for the longitudinally correlated nature of repeat measurements within a patient. Estimated mean changes and associated 90% confidence intervals will be reported. Primary secondary outcome is changes in weight.
Ambulatory activity levels | baseline, pre-intervention and immediately after the intervention
  Will be assessed by the within patient change in average daily steps taken within a week will be assessed from pre- to post-intervention. Mixed effects regression models will be used to estimate changes in ambulatory activity levels. Random effects will be included to account for the longitudinally correlated nature of repeat measurements within a patient. Estimated mean and associated 90% confidence interval will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Gorzelitz, PhD, Principal Investigator — University of Iowa Holden Comprehensive Cancer Center
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No